CLINICAL TRIAL: NCT06362187
Title: A Feasibility Study on Gut-Directed Virtual Reality for Chronic Pain Related to Chronic Pancreatitis
Brief Title: VR Pilot for Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Pandol, MD, Director, Basic and Translational Pancreas Research Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00003238
Record Dates: First submitted 2024-03-15; First posted 2024-04-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pancreatitis; Recurrent Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Gut Directed VR (Experimental)
  Interventions: Device: Gut Directed VR
- Sham VR (Sham Comparator)
  Interventions: Device: Sham Control VR

INTERVENTIONS:
Device: Gut Directed VR — The VR experiences follow a protocolized gut-directed therapy
  Arms: Gut Directed VR
Device: Sham Control VR — The same Oculus Quest 2 device as the active treatment group but will use distractive therapy
  Arms: Sham VR

SUMMARY:
The purpose of the research is to test the feasibility and preliminary impact of a home-based, standardized, gut-directed, virtual reality cognitive behavioral therapy (VR CBT) on clinical and functional outcomes of patients with chronic pancreatitis (CP) pain. The primary research procedures are questionnaires and biometric Fitbit data. The study will enroll adult patients with CP.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is a progressive inflammatory disease of the pancreas leading to fibrosis and permanent functional damage and associated with decreased health-related quality of life (HRQoL), impaired physical function, and frequent hospitalizations. Specifically, patients with CP often suffer from severe pain that impacts physical, social, and emotional wellbeing and leads to lost work productivity. Despite the substantial burden of pain, available therapies are limited in their ability to offer safe and effective analgesia. Although a stepwise approach has been applied to pain management, patients frequently turn to opioids, which can be associated with serious consequences including narcotic bowel syndrome and opioid-induced hyperalgesia. Hence, there is a critical gap in managing pain associated with CP.

Therapeutic virtual reality (VR) has emerged as an evidence-based, drug-free, immersive digital technology with established benefits for managing cognitive, affective, and sensory aspects of chronic pain. Unlike other audiovisual technologies, VR is in its ability to generate meaningful emotional experiences. Users of VR wear a head-mounted display that creates a vivid perception of being transported into immersive and emotionally evocative worlds. By stimulating the visual cortex while engaging other senses, VR distracts users from processing nociceptive stimuli while leveraging principles of CBT to enhance attitudes, beliefs, and cognitions about pain in a durable manner that does not require persistent use of VR once cognitive skills are transferred. Notably, in November of 2021, the U.S. Food and Drug Administration (FDA) authorized a CBT-based, 8-week, VR treatment course for chronic pain, supported by clinical trials from our team and others revealing evidence of clinical benefits.

Research indicates that VR offers clinical benefits for a variety of GI conditions including disorders of gut-brain interaction, perianal abscesses, sphincter of Oddi dysfunction. Previously, behavioral interventions such as CBT was emphasized by the International Consensus Guidelines for Chronic Pancreatitis in treating CP related pain when patients experience psychological impact of pain and quality of life has decreased. However, there are no existing study examining whether the benefits of therapeutic VR can also improve psychometric, biometric, and other clinical outcomes in CP patients.

This study aims to determine the feasibility of a home-based, standardized, gut-directed, VR CBT for patients with CP pain as well as investigate the preliminary impact of a home-based, standardized, gut-directed, VR CBT on clinical and functional outcomes of patients with CP pain. The study will also aim to isolate the immersive effect of gut-directed VR by comparing it with a non-immersive sham VR for patients with CP pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP [as determined by Cambridge 3-4 imaging classification (using CT, MRI, or MRCP) or a histologic diagnosis of CP]
* Clinically significant abdominal pain, measured using the standardized NIH PROMIS GI Pain Scale14 and defined as scoring at least 5 points above the nationally normed score (0.5 SD effect size), indicating equal or greater than the minimally clinically important difference (MCID) of abdominal pain
* Are 18-75 years of age
* Are able to read/write English. The study does not include non-English speakers as to current study material are only available in English.

Exclusion Criteria:

* Patients who are presenting with a condition that interferes with VR usage (e.g., seizures, facial injury precluding safe placement of headset, visual impairment)
* Patients who have cognitive impairment that affects protocol participation
* Patients who are recommended for long-term hospitalization
* Patients who are estimated to live <3 months from the time of enrollment
* Patients who have been diagnosed with a pancreatic tumor
* Patients who have been enrolled in an interventional/therapeutic drug trial for chronic or recurrent pancreatitis within the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of home-based VR | End of study (8 Weeks)
  The primary objective of this study is to determine the feasibility of a home-based, standardized, gut-directed, virtual reality cognitive behavioral therapy (VR CBT) on clinical and functional outcomes of patients with chronic pain from chronic pancreatitis (CP) based on subject's ability to adhere to and complete the study.
  Feasibility will be met if ≥75% of enrolled patients complete the 8-week study.

SECONDARY OUTCOMES:
Impact of home-based VR | End of study (8 Weeks)
  The secondary objective of this study is to investigate the preliminary impact of a home-based, standardized, gut-directed, VR CBT on clinical and functional outcomes of patients with CP pain.
  Health-related quality of life measurements will be collected via questionnaires to assess overall health, quality of life, and pain. An Acceptability Form will be provided during the last visit to gauge the general acceptability of the intervention. This data will be compared with biometric data obtained from a Fitbit device, including step counts, heart rate, and sleep parameters to assess the impact of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States